CLINICAL TRIAL: NCT05770245
Title: A Novel Electrolyzed Water Spray Reduces the Discomfort or Itching Scores, and Promotes Healing of the Damaged Skin of Patients With Mild Dermatophytosis: A Clinical Study
Brief Title: Novel Electrolyzed Water Spray Treatment Mild Dermatophytosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dove Medical Press Ltd (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: jia19650225
Record Dates: First submitted 2023-02-27; First posted 2023-03-15 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2023-02

CONDITIONS: Dermatophytoses
Keywords: Electrolyzed water device; Hydroxyl radical; Tap water; Spray; Dermatophytosis; Itching
MeSH Terms: conditions — Tinea; Pruritus

STUDY DESIGN:
Masking Description: An open label, single arm and before and after treatment comparison study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mild dermatophytosis and one treatment (Experimental): Study staff will use the novel electrolyzed water spray device and spray for approximately 10 minutes on the participant's diseased area until half a bottle (200ml) of water is used.
  Interventions: Device: The novel electrolyzed water spray

INTERVENTIONS:
Device: The novel electrolyzed water spray — The researcher used electrolyzed water or piped water to treat the diseased area two times a day for five days. The trial consists of 7 study visits (day 1-day 7). The reduction in the disease area of discomfort or itching scores and promoting healing of the damaged skin of patients with mild dermatophytosis event assessments will be performed at each visit. Safety analysis will be assessed based on the reports of adverse events during the study.

SUMMARY:
The purpose of this study is to test whether spraying the skin of patients of patients by use of the novel electrolyzed water spray will produce improvement in the condition of mild dermatophytosis.

DETAILED DESCRIPTION:
In this study, water inculding tap water,pure water and salt water, and an apparatus for producing electrolyzed water (https://www.deposon.com.cn; https://www.deposon.com）were used to generate an electrolyzed water mist spray or spray. This instantly generated electrolyzed water mist spray or spray has oxidation-reduction potential (ORP) ≥1200mv,and contains non-specific total oxidation capacity which equals to 0.28±0.10ppm,0.06±0.04ppm and 3.92±0.39ppm of desolved ozone. This instantly generated electrolyzed water mist spray or spray does not release detectable ≥0.1mg/m3 of gaseous ozone. This instantly generated electrolyzed water mist spray or spray has pH 8.4±0.4 and releases negative air ion.The apparatus for producing electrolyzed water has a positive electrode which is covered by a conductive diamond material (Patent# CN215308550U).This is an open-label, single-arm, and before and after treatment comparison study. This study uses this novel electrolyzed water device and the water spray to treat mild dermatophytosis.

ELIGIBILITY:
Inclusion Criteria:

* mild dermatophytosis accompanied by significant itching symptom
* Patient > 18 years old.

Exclusion Criteria:

* severe dermatophytosis.
* 80 years or older.
* Pregnant or breastfeeding women.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
An itching scale made by modifying the Numeric Pain Rating Scale (NPRS) | 7 days
  This Score is based on descriptions of the itching that patients rate 0-10 to assess the condition of their mild dermatophytosis. A higher score means a worse outcome. 0 means "no itching " and 10 means "the most itching".

SECONDARY OUTCOMES:
A skin signs scale made by modifying the Numeric Pain Rating Scale (NPRS). | 7 days
  The skin signs scale evaluates the disease-damaged skin replaced by fresh and healthy skin. This Score is based on descriptions of darkness or redness, swelling and dryness, broken surface, and reduced diseased skin area patients rate 0-10. A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Huinuode Biotechnology Co., Ltd., Qingdao, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: until publication of this clinical study and international patent granted